CLINICAL TRIAL: NCT00944255
Title: Pharmacogenetics of Antifolate Drugs in Autoimmune Diseases in Taiwan
Status: Completed | Type: Observational
Sponsor: National Chung Hsing University (Other)
Other Study IDs: C06289
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- RA with drug
- RA without drug

SUMMARY:
BACKGROUND. Polymorphisms occur in several genes encoding key enzymes in the folate pathway may affect drug metabolism in patients with rheumatoid arthritis. Whether these genetic variations contribute to differential responses to antifolate drug in patients with rheumatoid arthritis (RA) remains to be investigated in the Taiwanese population.

OBJECTIVE. The goal of the present study is to investigate the interactions between genetic variations in folate genes and the efficacy/side effects of anti-folate disease-modifying anti-rheumatic drug in Taiwan.

DESIGN. A cross-sectional study involving patients with RA were enrolled from TCVGH. Disease activity, drug efficacy and associated side-effects were assessed.

Genotypes in folylpoly-gamma-glutamate synthetase and reduced folate carrier were determined by RFLP or pyrosequencing.

ELIGIBILITY:
Inclusion Criteria:

* Male/female age >18
* RA diagnosed

Exclusion Criteria:

* Must not be pregnant/breastfeeding
* Other conditions may lead to exclusion from the trial (e.g. Diabetes mellitus, malignant melanoma, cardiac conduction disorders, hepatic/renal insufficiency.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cross-sectional study involving 150 patients with RA were enrolled from TCVGH.
Sampling Method: Probability Sample
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)